CLINICAL TRIAL: NCT02833987
Title: The Comparative Safety of Direct Oral Anticoagulants Versus Warfarin for the Treatment of Venous Thromboembolism
Brief Title: Direct Oral Anticoagulants and Venous Thromboembolism
Status: Completed | Type: Observational
Sponsor: Canadian Network for Observational Drug Effect Studies, CNODES (Other)
Collaborators: Drug Safety and Effectiveness Network, Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: Q14-02
Record Dates: First submitted 2016-07-11; First posted 2016-07-15 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Venous Thromboembolism; Major Bleed
Keywords: Direct oral anticoagulants; Safety; Major bleed; Adverse events
MeSH Terms: conditions — Venous Thromboembolism | interventions — apixaban; Dabigatran; Rivaroxaban; Warfarin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Treated with direct oral anticoagulants (DOACs): Patients who received a new prescription for a DOAC (apixaban, dabigatran, or rivaroxaban) in the 30 days following the date of an incident VTE diagnosis, and did not have a previous prescription for a DOAC or warfarin in the year prior to the date of the new prescription.
  Interventions: Drug: Apixaban (ATC B01AF02); Drug: Dabigatran (ATC B01AE07); Drug: Rivaroxaban (ATC B01AF01)
- Treated with warfarin: Patients who received a new prescription for warfarin in the 30 days following the date of an incident VTE diagnosis, and did not have a previous prescription for a DOAC or warfarin in the year prior to the date of the new prescription.
  Interventions: Drug: Warfarin (ATC B01AA03)

INTERVENTIONS:
Drug: Apixaban (ATC B01AF02) — Exposure to apixaban (ATC B01AF02) will be defined as a new prescription for apixaban in the 30 days following the date of an incident VTE diagnosis.
  Groups: Treated with direct oral anticoagulants (DOACs)
Drug: Dabigatran (ATC B01AE07) — Exposure to dabigatran (ATC B01AE07) will be defined as a new prescription for dabigatran in the 30 days following the date of an incident VTE diagnosis.
  Groups: Treated with direct oral anticoagulants (DOACs)
Drug: Rivaroxaban (ATC B01AF01) — Exposure to rivaroxaban (ATC B01AF01) will be defined as a new prescription for rivaroxaban in the 30 days following the date of an incident VTE diagnosis.
  Groups: Treated with direct oral anticoagulants (DOACs)
Drug: Warfarin (ATC B01AA03) — Exposure to warfarin (ATC B01AA03) will be defined as a new prescription for warfarin in the 30 days following the date of an incident VTE diagnosis.
  Groups: Treated with warfarin

SUMMARY:
The purpose of this study is to determine whether use of direct oral anticoagulants (DOACs) is associated with an increased risk of major bleeding compared to warfarin use, for the treatment of venous thromboembolism (VTE).

The investigators will carry out separate population based cohort studies using health administrative databases in eight jurisdictions in Canada, the UK and the US. Cohorts will be defined by the initiation of a DOAC or warfarin on or after January 1, 2009, with an incident diagnosis of VTE having occurred within 30 days prior to the date of the prescription for the DOAC or warfarin. Follow-up will continue until a hospitalization or emergency department visit for a major bleed. The results from separate sites will be combined to provide an overall assessment of the risk of major bleeding in DOAC users.

DETAILED DESCRIPTION:
The objective of this study is to determine whether the use of direct oral anticoagulants (DOACs) is associated with an increased risk of major bleeding compared to warfarin use, for the treatment of venous thromboembolism (VTE).

A common-protocol approach will be used to conduct retrospective cohort studies using administrative health care data from eight jurisdictions (the Canadian provinces of Alberta, Manitoba, Nova Scotia, Ontario, Quebec, Saskatchewan, as well as the United Kingdon (UK) Clinical Practice Research Datalink and the United States (US) Marketscan). Briefly, the Canadian databases include population-level data on physician billing, diagnoses and procedures from hospital discharge abstracts, and dispensations for prescription drugs. The data in Nova Scotia, Ontario, and Alberta will be restricted to patients aged 65 years and older, as prescription data are not available for younger patients. The CPRD is a clinical database that is representative of the UK population and contains the records for patients seen at over 680 general practitioner practices in the UK.

In each jurisdiction, the investigators will assemble a study cohort that includes all patients newly prescribed a DOAC or warfarin from January 1, 2009 (or the earliest date of data availability at each site) to October 2, 2014 (or 180 days before the last date of data availability at each site, if earlier), that had an incident diagnosis of VTE within the 30 days prior to the date of the prescription. The date of study cohort entry will be defined by the prescription (for CPRD) or dispensation (for all other sites) date of the newly prescribed DOAC or warfarin. Patients in the study cohort will be followed from the date of study cohort entry until an event (defined below), censoring due to death or departure from the database, 3 months after cohort entry, or the end of the study period (March 31, 2015), whichever occurs first.

Exposure to a DOAC will be defined as a new prescription for a DOAC on the date of cohort entry. Exposure to warfarin will be defined as a new prescription for warfarin on the date of cohort entry. The investigators will use an analysis analogous to an intention-to-treat approach. The primary outcome will be defined as a hospitalization or emergency department visit for a major bleed within 3 months of cohort entry.

The study cohort will be analyzed using a matched cohort design, where up to 5 warfarin users will be matched to each DOAC user on sex, age, cohort entry date, and propensity score (which will be constructed using a multivariable logistic regression model estimating the odds of being treated with DOACs, while adjusting for a number of pre-identified covariates to account for baseline difference at the time of cohort entry). The hazard of major bleeding with DOAC use vs. warfarin use will be estimated using Cox-proportional hazards regression models accounting for the potential correlation in the matched pairs. Meta-analyses of the site-specific results will then be performed using fixed or random effects models (according to results of Chi-squared tests for heterogeneity). Sensitivity analyses will be conducted, all defined a priori, to assess the robustness of the results.

As secondary analyses, the investigators will: 1) assess the risk of all-cause mortality associated with DOAC use compared to warfarin use in the 3 months after cohort entry; 2) assess the risk of major bleeding associated with DOAC use compared to warfarin use, according to chronic kidney disease status; 3) determine (descriptively) the proportion of patients who experienced a major bleeding event by major bleed type; and 4) stratify the primary analysis by age (less than 66, 66-75, 76-85 and greater than 85), sex, and use of an anti-platelet medication in the 90 day period prior to cohort entry.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a new prescription for a DOAC or warfarin that had an incident diagnosis of VTE within the 30 days prior to the date of the prescription
* Patients at least 18 years of age (except Nova Scotia, Ontario, and Alberta, where patients will be at least 66 years of age)
* Patients with at least 1 year of history in the database

Exclusion Criteria:

* Patients with a diagnosis of VTE or atrial fibrillation ≤335 days prior to the incident VTE diagnosis
* Patients that received a prescription for a DOAC or warfarin within 1 year prior to the date of the cohort entry
* Patients who received prescriptions for both a DOAC and warfarin on the date of cohort entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In each jurisdiction, the investigators will assemble a study cohort that includes all patients aged 18 years or older with a new prescription for a DOAC or warfarin between January 1, 2009 and 180 days prior to the end date of data availability within that jurisdiction and with an incident diagnosis of VTE within 30 days prior to the date of the cohort entry prescription.
Sampling Method: Probability Sample
Enrollment: 59525 (Actual)
Dates: Start 2015-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Major bleed | Patients will be followed from the date of the first DOAC or warfarin prescription (study cohort entry) to a hospitalization or emergency department visit for a major bleed, censoring, or for up to 3 months, whichever occurred first.
  Patients hospitalized or visiting the emergency department for a major bleed recorded as the most responsible diagnosis in either the discharge abstract or hospitalization record with the following ICD codes:
  ICD-9 codes: 430, 431, 432.0, 432.1, 432.9, 531.0, 531.2, 531.4, 531.6, 532.0, 532.2, 532.4, 532.6, 533.0, 533.2, 533.4, 533.6, 534.0, 534.2, 534.4, 534.6, 578.0, 578.1, 578.9, 569.3, 578.1, 578.9
  ICD-10 codes: I60, I61, I62.0, I62.1, I62.9, K92.0, K92.1, I85.0, I98.20, I98.3, K22.10, K22.12, K22.14, K22.16, K25.0, K25.2, K25.4, K25.6, K26.0, K26.2, K26.4, K26.6, K27.0, K27.2, K27.4, K27.6, K28.0, K28.2, K28.4, K28.6, K29.0, K63.80, K31.80, K55.20, K62.5, K92.2, N02.0, N02.1, N02.2, N02.3, N02.4, N02.5, N02.6, N02.7, N02.8, N02.9, K66.1, N93.8, N93.9, N95.0, R04.1, R04.2, R04.8, R04.9, R31.0, R31.1, R31.8, R58, D68.3, H35.6, H43.1, H45.0, M25.0

SECONDARY OUTCOMES:
All-cause mortality | Patients were followed from the date of the first DOAC or warfarin prescription (study cohort entry) until death, censoring or for up to 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Hemmelgarn, MD, PhD, Principal Investigator — Department of Community Health Sciences, University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Result] Jun M, Lix LM, Durand M, Dahl M, Paterson JM, Dormuth CR, Ernst P, Yao S, Renoux C, Tamim H, Wu C, Mahmud SM, Hemmelgarn BR; Canadian Network for Observational Drug Effect Studies (CNODES) Investigators. Comparative safety of direct oral anticoagulants and warfarin in venous thromboembolism: multicentre, population based, observational study. BMJ. 2017 Oct 17;359:j4323. doi: 10.1136/bmj.j4323. PMID 29042362
- See also: This organization's website describing general functions, other CNODES projects, and investigator profiles. — http://www.cnodes.ca